CLINICAL TRIAL: NCT01092416
Title: Pivotal Trial to Evaluate the Safety and Efficacy of the Diamondback 360°® Orbital Atherectomy System in Treating De Novo, Severely Calcified Coronary Lesions (ORBIT II)
Brief Title: Evaluate the Safety and Efficacy of OAS in Treating Severely Calcified Coronary Lesions
Acronym: ORBIT II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORBIT II
Record Dates: First submitted 2010-03-23; First posted 2010-03-25 (Estimated); Results first posted 2016-01-06 (Estimated); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Coronary Artery Disease
Keywords: CAD; Severely calcified lesion
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Diamondback 360 Orbital Atherectomy System — Diamondback 360 Orbital Atherectomy System. The (OAS) utilizes a diamond-coated eccentric crown that, while rotating over an atherectomy guide wire, expands the lumen diameter laterally via centrifugal forces (up to a maximum orbit diameter for a given rotational speed and crown diameter). It is a minimally invasive PCI procedure.

SUMMARY:
This is a prospective, single-arm, multi-center study to evaluate the safety and performance of the OAS in treating de novo, severely calcified coronary lesions in adult subjects. Study is going to enroll up to 429 subjects in up to 50 U.S. study sites. The primary safety endpoint is 30-day MACE and primary efficacy endpoint is procedural success. All subjects will be treated with the orbital atherectomy system and adjunctive stent. All subjects will be followed in clinic at 30 days. Additionally, all subjects will have an annual phone call or clinical follow up at each anniversary until study is closed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 or older.
* Subjects must have a clinical indication for coronary intervention.
* CK and CK-MB must be less than or equal to the upper limit of lab normal value within 8 hours prior to the procedure.
* The target lesion must be a de novo coronary lesion that has not been previously treated with any interventional procedure.
* The target vessel must be a native coronary artery with a stenosis of >= 70% and < 100%.
* The target vessel reference diameter must be >= 2.5mm and <= 4.0 mm.
* The lesion length must not exceed 40 mm.
* The target vessel must have a TIMI flow 3 at baseline.
* The target lesion must have evidence of severe calcium deposit at the lesion site based on the protocol criterion.
* The lesion must be crossable with the study guide wire.

Exclusion Criteria:

* Inability to understand the study or a history of non-compliance with medical advice.
* Unwilling or unable to sign the ORBIT II Informed Consent Form (ICF).
* History of any cognitive or mental health status that would interfere with study participation.
* Currently enrolled in any other pre-approval investigational study (does not apply to long-term post-market studies unless these studies might clinically interfere with the current study endpoints (e.g., limit use of study-required medication, etc.).
* Female subjects who are pregnant or planning to become pregnant within the study period.
* Known hypersensitivity or contraindication to aspirin, heparin, ticlopidine or clopidogrel without adequate alternative medications.
* Known sensitivity to contrast media, which cannot be adequately pre-medicated.
* Diagnosed with chronic renal failure or has a serum creatinine level >2.5 mg/dl.
* Experienced acute MI (STEMI or non-STEMI: CK and CK-MB greater than 1 times the upper limit of lab normal) within 30 days prior to index procedure.
* History of major cardiovascular intervention within 30 days.
* Evidence of current (within 6 months) left ventricular ejection fraction ≤ 25%.
* NYHA class III or IV heart failure.
* History of a stroke or transient ischemic attack (TIA) within 6 months.
* Active peptic ulcer or upper gastrointestinal (GI) bleeding within 6 months.
* History of bleeding diathesis or coagulopathy or intention to refuse blood transfusion if one should become necessary.
* Concurrent medical condition with a life expectancy of less than 12 months.
* History of immune deficiency.
* Uncontrolled insulin dependent diabetes.
* Evidence of active infections on the day of the index procedure.
* Subject has planned cardiovascular intervention within 60-days post index procedure.
* Subject is not an acceptable candidate for emergent coronary artery bypass surgery.
* Subject with known allergy to atherectomy lubricant components such as soybean oil, egg yolk phospholipids, glycerin and sodium hydroxide.
* Subject with 3 lesions requiring intervention.
* Subject with 2 lesions unless the treatment of the lesions is staged. The non target lesion must first be treated at least 12 hours prior to the index procedure. The subject's CK and CK-MB must be less than or equal to one times the upper limit of the lab normal value 12 ± 2 hours post procedure and there were no procedural complications during the first lesion intervention.
* Target lesion is located in a native vessel distal to anastomosis with a saphenous vein graft or LIMA/RIMA bypass.
* Target vessel has other lesions with greater than 50% diameter stenosis based on visual estimate or on-line QCA.
* Target vessel has angiographically visible or suspected thrombus.
* Target vessel has a stent from previous PCI.
* Target vessel is excessively tortuous.
* Target lesion is an ostial location (within 5 mm of ostium) or an unprotected left main lesion.
* Target lesion is a bifurcation.
* Target lesion has a ≥ 1.5 mm side branch.
* Angiographic evidence of a dissection prior to OAS treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 443 (Actual)
Dates: Start 2010-05; Primary Completion 2013-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Chambers, MD, Principal Investigator — Metropolitan Cardiology Consutants
Locations (51):
- United States (51):
  - Trinity Hospital, Birmingham, Alabama
  - Baptist Montgomery South, Montgomery, Alabama
  - Mercy Gilbert, Gilbert, Arizona
  - Cedar Sinai Los Angeles, Beverly Hills, California
  - Good Samaritan Hospital, Los Angeles, California
  - Eisenhower Medical Center, Palm Springs, California
  - Desert Cardiology Center, Rancho Mirage, California
  - Sutter Memorial Hospital, Sacramento, California
  - Florida Hospital Memorial, Daytona Beach, Florida
  - North Florida Regional, Gainesville, Florida
  - Munroe Regional Medical Center, Ocala, Florida
  - Florida Hospital, Orlando, Florida
  - Orlando Regional, Orlando, Florida
  - Palm Beach Gardens, Palm Beach Gardens, Florida
  - Winter Haven, Winter Haven, Florida
  - Emory University, Atlanta, Georgia
  - Indiana Heart Hospital, Indianapolis, Indiana
  - Saint Vincents Indianapolis, Indianapolis, Indiana
  - Community Hospital, Munster, Indiana
  - Iowa Heart, Des Moines, Iowa
  - Kansas University Medical Center, Kansas City, Kansas
  - King's Daughters / Kentucky Heart Foundation, Ashland, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Cape Cod Research Institute, Hyannis, Massachusetts
  - Detroit Medical Center, Detroit, Michigan
  - St. John's Hospital, Detroit, Michigan
  - St. Joseph Mercy, Pontiac, Michigan
  - Lakeland, Saint Joseph, Michigan
  - Mercy Hospital, Coon Rapids, Minnesota
  - Abbott Northwestern, Minneapolis, Minnesota
  - United Heart & Vascular, Saint Paul, Minnesota
  - North Mississippi Medical Center, Tupelo, Mississippi
  - Saint Michaels, Newark, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - New York Methodist Hospital, Brooklyn, New York
  - Columbia University Medical Center, New York, New York
  - Lenox Hill, New York, New York
  - St. Francis, Roslyn, New York
  - Good Samaritan Dayton, Dayton, Ohio
  - Oklahoma Heart, Oklahoma City, Oklahoma
  - The Heart and Vascular Center, Beaver, Pennsylvania
  - Bryn Mawr / Lankenau, Bryn Mawr, Pennsylvania
  - St. Mary's, Langhorne, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Baptist Memorial Hospital-DeSoto, Memphis, Tennessee
  - Baylor, Dallas, Texas
  - Memorial Hermann, Houston, Texas
  - St. Luke's, Houston, Texas
  - Davis Hospital, Layton, Utah
  - Saint Joe Bellingham / North Cascade Cardiology, Bellingham, Washington

REFERENCES:
- [Result] Genereux P, Lee AC, Kim CY, Lee M, Shlofmitz R, Moses JW, Stone GW, Chambers JW. Orbital Atherectomy for Treating De Novo Severely Calcified Coronary Narrowing (1-Year Results from the Pivotal ORBIT II Trial). Am J Cardiol. 2015 Jun 15;115(12):1685-90. doi: 10.1016/j.amjcard.2015.03.009. Epub 2015 Mar 24. PMID 25910525
- [Result] Chambers JW, Feldman RL, Himmelstein SI, Bhatheja R, Villa AE, Strickman NE, Shlofmitz RA, Dulas DD, Arab D, Khanna PK, Lee AC, Ghali MG, Shah RR, Davis TP, Kim CY, Tai Z, Patel KC, Puma JA, Makam P, Bertolet BD, Nseir GY. Pivotal trial to evaluate the safety and efficacy of the orbital atherectomy system in treating de novo, severely calcified coronary lesions (ORBIT II). JACC Cardiovasc Interv. 2014 May;7(5):510-8. doi: 10.1016/j.jcin.2014.01.158. PMID 24852804
- [Result] Lee M, Genereux P, Shlofmitz R, Phillipson D, Anose BM, Martinsen BJ, Himmelstein SI, Chambers JW. Orbital atherectomy for treating de novo, severely calcified coronary lesions: 3-year results of the pivotal ORBIT II trial. Cardiovasc Revasc Med. 2017 Jun;18(4):261-264. doi: 10.1016/j.carrev.2017.01.011. Epub 2017 Jan 23. PMID 28162989
- [Result] Genereux P, Bettinger N, Redfors B, Lee AC, Kim CY, Lee MS, Shlofmitz RA, Moses JW, Stone GW, Chambers JW. Two-year outcomes after treatment of severely calcified coronary lesions with the orbital atherectomy system and the impact of stent types: Insight from the ORBIT II trial. Catheter Cardiovasc Interv. 2016 Sep;88(3):369-77. doi: 10.1002/ccd.26554. Epub 2016 Apr 16. PMID 27084293
- [Result] Shlofmitz E, Martinsen BJ, Behrens AN, Ali ZA, Lee MS, Puma JA, Shlofmitz RA, Chambers JW. Direct Stenting in Patients Treated with Orbital Atherectomy: An ORBIT II Subanalysis. Cardiovasc Revasc Med. 2019 Jun;20(6):454-460. doi: 10.1016/j.carrev.2019.03.011. Epub 2019 Mar 21. PMID 30982659
- [Result] Lee MS, Shlofmitz RA, Shlofmitz E, Behrens AN, Revtyak G, Martinsen BJ, Chambers JW. Procedural and Long-Term Ischemic Outcomes of Tight Subtotal Occlusions Treated with Orbital Atherectomy: An ORBIT II Subanalysis. Cardiovasc Revasc Med. 2019 Jul;20(7):563-568. doi: 10.1016/j.carrev.2018.09.011. Epub 2018 Sep 13. PMID 30243964
- [Result] Lee MS, Shlofmitz RA, Shlofmitz E, Srivastava PK, Kong J, Grines C, Revytak G, Chambers JW. Orbital atherectomy for the treatment of small (2.5mm) severely calcified coronary lesions: ORBIT II sub-analysis. Cardiovasc Revasc Med. 2018 Apr;19(3 Pt A):268-272. doi: 10.1016/j.carrev.2017.09.017. Epub 2017 Oct 3. PMID 29454531
- [Result] Lee MS, Shlofmitz RA, Martinsen BJ, Sethi S, Chambers JW. Impact of age following treatment of severely calcified coronary lesions with the orbital atherectomy system: 3-year follow-up. Cardiovasc Revasc Med. 2018 Sep;19(6):655-659. doi: 10.1016/j.carrev.2018.01.011. Epub 2018 Jan 31. PMID 29452841
- [Result] Lee MS, Anose BM, Martinsen BJ, Lee AC, Shlofmitz RA, Chambers JW. Orbital atherectomy treatment of severely calcified native coronary lesions in patients with prior coronary artery bypass grafting: Acute and one-year outcomes from the ORBIT II trial. Cardiovasc Revasc Med. 2018 Jul;19(5 Pt A):498-502. doi: 10.1016/j.carrev.2017.10.009. Epub 2017 Nov 5. PMID 29117920
- [Result] Shlofmitz E, Martinsen B, Lee M, Genereux P, Behrens A, Kumar G, Puma J, Shlofmitz R, Chambers J. Utilizing intravascular ultrasound imaging prior to treatment of severely calcified coronary lesions with orbital atherectomy: An ORBIT II sub-analysis. J Interv Cardiol. 2017 Dec;30(6):570-576. doi: 10.1111/joic.12423. Epub 2017 Aug 7. PMID 28786143
- [Result] Lee MS, Martinsen BJ, Lee AC, Behrens AN, Shlofmitz RA, Kim CY, Chambers JW. Impact of diabetes mellitus on procedural and one year clinical outcomes following treatment of severely calcified coronary lesions with the orbital atherectomy system: A subanalysis of the ORBIT II study. Catheter Cardiovasc Interv. 2018 May 1;91(6):1018-1025. doi: 10.1002/ccd.27208. Epub 2017 Jul 22. PMID 28733974
- [Result] Lee MS, Martinsen BJ, Shlofmitz R, Shlofmitz E, Lee AC, Chambers J. Orbital atherectomy treatment of severely calcified coronary lesions in patients with impaired left ventricular ejection fraction: one-year outcomes from the ORBIT II study. EuroIntervention. 2017 Jun 20;13(3):329-337. doi: 10.4244/EIJ-D-16-00301. PMID 28191873
- [Result] Lee MS, Lee AC, Shlofmitz RA, Martinsen BJ, Hargus NJ, Elder MD, Genereux P, Chambers JW. ORBIT II sub-analysis: Impact of impaired renal function following treatment of severely calcified coronary lesions with the Orbital Atherectomy System. Catheter Cardiovasc Interv. 2017 Apr;89(5):841-848. doi: 10.1002/ccd.26778. Epub 2016 Aug 27. PMID 27567020
- [Result] Lee MS, Shlofmitz E, Shlofmitz R, Sahni S, Martinsen B, Chambers J. Outcomes After Orbital Atherectomy of Severely Calcified Left Main Lesions: Analysis of the ORBIT II Study. J Invasive Cardiol. 2016 Sep;28(9):364-9. Epub 2016 Mar 15. PMID 26984932
- [Result] Kim CY, Lee AC, Wiedenbeck TL, Lee MS, Chambers JW. Gender differences in acute and 30-day outcomes after orbital atherectomy treatment of de novo, severely calcified coronary lesions. Catheter Cardiovasc Interv. 2016 Mar;87(4):671-7. doi: 10.1002/ccd.26163. Epub 2015 Sep 2. PMID 26331279

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study received approval to enroll up to 429 subjects. Following the introduction of the Electric OAS, the enrollment was expanded to a maximum of 479 subjects, to enroll 100 subjects with the Electric OAS. A total of 443 subjects were enrolled in the study between May 25, 2010 and November 26, 2012 at 49 U.S. study sites.
Pre-assignment Details: A subject was considered enrolled when a signed informed consent was in place, all inclusion/no exclusion criteria were met, and the study guidewire had crossed the target lesion.
Groups:
- ORBIT II Subjects: Subjects enrolled in ORBIT II study.
Period: Enrollment
Arm/Group | ORBIT II Subjects
Started | 443
Completed | 440
Not Completed | 3
Not completed — Atherectomy device not inserted | 3
Period: 30-Day Follow-up
Arm/Group | ORBIT II Subjects
Started | 440
Completed | 430
Not Completed | 10
Not completed — Death | 2
Not completed — Missed 30-day follow-up | 3
Not completed — Data collected after close of 30D window | 5
Period: 12-Month Follow-up
Arm/Group | ORBIT II Subjects
Started | 438
Completed | 413
Not Completed | 25
Not completed — Death | 16
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 2
Not completed — Missed 1-year follow-up | 1
Not completed — Data collected after close of 1Y window | 2

BASELINE CHARACTERISTICS:
Arm/Group | ORBIT II Subjects
Number analyzed (Participants) | 443
Age, Continuous [Mean (Full Range); unit: years] | 71.4 [37.4 to 92.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 157
  Male | 286
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 390
  Black or African American | 25
  Asian | 9
  Hispanic or Latino | 15
  Native American | 1
  Other | 3

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint: 30-Day Freedom From Major Adverse Cardiac Events (MACE)
Description: OAS safety was measured by a composite of MACE at 30-days post procedure. MACE is composed of:
  * Cardiac death.
  * MI - defined as a CK-MB level > 3 times the upper limit of lab normal (ULN) value with or without new pathologic Q wave.
  * TVR - defined as revascularization at the target vessel (inclusive of the target lesion) after the completion of the index procedure.
Time Frame: 30 days
Population: A Kaplan-Meier analysis was performed to determine the percent probability that a study participant is free from major adverse cardiac events at 30 days.
Measure: Number (95% Confidence Interval); unit: Percent probability of Freedom from MACE
Arm/Group | ORBIT II Subjects
Number analyzed (Participants) | 443
Percent probability of Freedom from MACE | 89.6 [86.7 to 92.5]

2. Secondary Outcome: Angiographic Success
Description: Angiographic success was defined as success in facilitating stent delivery with <50% residual stenosis and without severe angiographic complications.
Time Frame: Baseline procedure, with a mean total procedure time of 52.5 minutes.
Measure: Number; unit: Percentage of procedures
Arm/Group | ORBIT II Subjects
Number analyzed (Participants) | 443
Percentage of procedures | 91.4

3. Secondary Outcome: Severe Angiographic Complications
Description: Severe angiographic complications were defined as severe dissection (Type C to F), perforation, abrupt closure, and persistent slow flow or persistent no reflow.
Time Frame: Baseline procedure, with a mean total procedure time of 52.5 minutes.
Measure: Number; unit: Participants
Arm/Group | ORBIT II Subjects
Number analyzed (Participants) | 443
Participants
  Type C, D, E, or F Dissection | 15
  Perforation | 8
  Persistent Slow Flow | 4
  Persistent No Reflow | 0
  Abrupt Closure | 8

4. Secondary Outcome: 12-Month Freedom From Major Adverse Cardiac Events (MACE)
Description: The safety of the OAS was measured for the secondary safety endpoint consisting of a composite of freedom from MACE through 12 months of follow-up.
Time Frame: 12 months
Population: A Kaplan-Meier analysis was performed to determine the percent probability that a study participant is free from major adverse cardiac events at 12 months.
Measure: Number (95% Confidence Interval); unit: Percent probability of Freedom from MACE
Arm/Group | ORBIT II Subjects
Number analyzed (Participants) | 443
Percent probability of Freedom from MACE | 83.1 [79.6 to 86.7]

5. Primary Outcome: Primary Efficacy Endpoint: Procedural Success
Description: Procedural success was defined as success in facilitating stent delivery with a residual stenosis of <50% and without the occurrence of an in-hospital MACE in de novo, severely calcified coronary lesions.
Time Frame: Participants were followed from baseline procedure through the duration of hospital stay, an average of 33.6 hours.
Measure: Number (95% Confidence Interval); unit: Percentage of procedures
Groups:
- OAS Treatment Group: Subjects enrolled in ORBIT II study and in whom the atherectomy device was inserted.
Arm/Group | OAS Treatment Group
Number analyzed (Participants) | 440
Percentage of procedures | 88.9 [85.5 to 91.6]

ADVERSE EVENTS:
Description: Serious Adverse Events reported by sites and adjudicated by the Clinical Events Committee.
Groups:
- ORBIT II Subjects - 30 Day Results: Serious Adverse Events reported out to 30 Days Post-Procedure for Subjects enrolled in ORBIT II study.
- ORBIT II Subjects - 1 Year Results: Serious Adverse Events reported from 31 Days to 1 Year Post-Procedure for Subjects enrolled in ORBIT II study.
Arm/Group | ORBIT II Subjects - 30 Day Results | ORBIT II Subjects - 1 Year Results
Serious Adverse Events (participants affected / at risk) | 109/443 | 70/438
Other Adverse Events (participants affected / at risk) | 34/443 | 0/438
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ORBIT II Subjects - 30 Day Results (N=443) | ORBIT II Subjects - 1 Year Results (N=438)
Acute MI, Q-wave (Cardiac disorders) | 4 (4) | 0 (0)
Acute MI, non Q-wave (Cardiac disorders) | 39 (39) | 5 (5)
Angina Pectoris (Cardiac disorders) | 4 (4) | 23 (25)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 9 (9)
Atrioventricular block, II degree (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac/pericardial tamponade (Cardiac disorders) | 4 (4) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 2 (2) | 0 (0)
Chest pain (Cardiac disorders) | 2 (2) | 3 (3)
Endocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Non-target vessel revascularization (Cardiac disorders) | 1 (1) | 3 (4)
PEA arrest (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Shock (Acute RV dysfunction and acute blood loss hypovolemic) (Cardiac disorders) | 1 (1) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 1 (1) | 2 (2)
Ventricular fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia/ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery embolism of air, plaque, thrombosis, or debris (Surgical and medical procedures) | 3 (3) | 0 (0)
Slow flow or no reflow phenomena (Surgical and medical procedures) | 3 (3) | 0 (0)
Thrombosis formation at site of treated lesion (Surgical and medical procedures) | 1 (1) | 0 (0)
Hematoma at access site, requiring intervention (Vascular disorders) | 1 (1) | 0 (0)
Hemorrhage, major, requiring transfusion (Vascular disorders) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 2 (2)
Peripheral artery pseudoaneurysm (Vascular disorders) | 3 (3) | 0 (0)
Peripheral artery/vascular disease (Vascular disorders) | 2 (2) | 9 (10)
Pulmonary embolism (Vascular disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (CVA) (Nervous system disorders) | 3 (3) | 2 (2)
Sundowning/ICU "psychosis" (Nervous system disorders) | 1 (1) | 0 (0)
Anoxia due to aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (14)
Dyspnea/Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (7)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6)
Respiratory failure, requiring intubation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 4 (4)
Esophageal spasm (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal bleeding (Gastrointestinal disorders) | 3 (3) | 5 (5)
Nausea and/or vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Renal insufficiency (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary tract infection (UTI) (Renal and urinary disorders) | 1 (1) | 5 (5)
Cardiac death (Cardiac disorders) | 1 (1) | 12 (12)
Non-cardiac death (General disorders) | 1 (1) | 4 (4)
Bone fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6)
Fever (General disorders) | 1 (1) | 0 (0)
Infection at access site (Infections and infestations) | 1 (1) | 0 (0)
Left arm AV graft infection (Infections and infestations) | 1 (1) | 0 (0)
Lower extremity pain (General disorders) | 1 (1) | 0 (0)
Coronary vessel dissection present (Surgical and medical procedures) | 23 (23) | 0 (0)
Coronary vessel perforation present (Surgical and medical procedures) | 8 (8) | 0 (0)
Non-coronary right ventricle vessel perforation present (Surgical and medical procedures) | 1 (1) | 0 (0)
Acute congestive heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 2 (2)
Arrhythmia, unspecified (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Chronic congestive heart failure, or exacerbation (Cardiac disorders) | 0 (0) | 8 (12)
Coronary artery restenosis (Cardiac disorders) | 0 (0) | 20 (22)
Heart flutter/nervous feeling in chest (Cardiac disorders) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Pacemaker end of life (Cardiac disorders) | 0 (0) | 1 (1)
Palpitation (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Carotid artery disease (Vascular disorders) | 0 (0) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Anxiety (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral artery aneurysm (Vascular disorders) | 0 (0) | 2 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Mental status changes (Nervous system disorders) | 0 (0) | 2 (2)
Panic attack (Nervous system disorders) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 8 (9)
Tinnitus (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischemic attack (TIA) (Nervous system disorders) | 0 (0) | 2 (2)
Vasovagal reaction (Nervous system disorders) | 0 (0) | 1 (1)
Flu (Infections and infestations) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Multiple lymphadenopathy (on chest CT) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory infection (Infections and infestations) | 0 (0) | 2 (2)
Bile duct leak (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biloma (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Complicated appendicitis (rupture) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Complications post cholecystectomy (Hepatobiliary disorders) | 0 (0) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Elevated liver function tests (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallstone (Hepatobiliary disorders) | 0 (0) | 2 (2)
Gangrenous gallbladder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 4 (4)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectocoele repair (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 0 (0) | 6 (6)
Chronic renal failure, or exacerbation (Renal and urinary disorders) | 0 (0) | 2 (2)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Obstructive uropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal calculi (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 5 (5)
Hyponatremia (General disorders) | 0 (0) | 1 (1)
Supratherapeutic INR (General disorders) | 0 (0) | 1 (1) — International Normalized Ratio/Prothrombin time
Death, unknown cause (General disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 9 (9)
Arthroplasty revision (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (General disorders) | 0 (0) | 1 (1)
Bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Bilateral cataracts (Eye disorders) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Carpal tunnel syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cellulitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Chest pain, non-cardiac (General disorders) | 0 (0) | 1 (1)
Epistaxis (General disorders) | 0 (0) | 1 (1)
Fall/Loss of balance (General disorders) | 0 (0) | 2 (2)
Gout (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Hernia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Infection at pacemaker site (Infections and infestations) | 0 (0) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Metabolic acidosis (General disorders) | 0 (0) | 2 (2)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Peripheral edema (General disorders) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gynecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Knee replacement (Surgical and medical procedures) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Spinal stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Trauma (General disorders) | 0 (0) | 3 (3)
Gangrene (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ORBIT II Subjects - 30 Day Results (N=443) | ORBIT II Subjects - 1 Year Results (N=438)
Angiographic Complications (Surgical and medical procedures) | 34 (34) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any previously unpublished information provided to the Investigators by the Sponsor is confidential and will remain the sole property of the Sponsor. The Investigator agrees to use this information only in accomplishing this study not use it for other purposes without the Sponsor's written consent. An Investigator can generate additional publication ideas based on the trial data. The Sponsor reserves the right to review the manuscript prior to submission in order to verify accuracy of the data.